CLINICAL TRIAL: NCT02351596
Title: The Effect of a 'Core Stability' Physiotherapy Group Intervention Programme on Balance in Ambulant Children With Cerebral Palsy: A Randomised Control Trial
Brief Title: Do Core Stability Exercise Classes Help Children With Cerebral Palsy Improve Their Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Central Remedial Clinic (Unknown)
Responsible Party: Principal Investigator, Dara Meldrum, Dr. Dara Meldrum BSc, MSc, PhD (NUI, RCSI), MISCP, Royal College of Surgeons, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPSP1415
Record Dates: First submitted 2014-12-10; First posted 2015-01-30 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Cerebral Palsy
Keywords: Core Stability; Balance; Core Control
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention Group 7-12 years (Active Comparator): Intervention consists of attending a Physiotherapy Core stability group programme for 8 sessions over 4 weeks. Each session lasts 60 minutes (mins).
  Dosage: 60minsX 2 =120mins/week X 4 = 480 mins total dosage of intervention Participants also given a home exercise programme with a diary to record how long they practice for every day.
  Interventions: Other: Physiotherapy Core Stability Group Programme
- Control Group 7-12 years (Active Comparator): Participants continue with usual care but do not include core stability or balance specific exercises in their physiotherapy programme for the duration of the control period. If they are receiving active physiotherapy treatment during this time, the duration, type and frequency of this intervention is recorded.
  Interventions: Other: Control Group
- Clontarf Intervention Group 13-17 years (Active Comparator): Intervention consists of attending a Physiotherapy Core stability group programme for 8 sessions over 4 weeks. Each session lasts 60 minutes (mins).
  Dosage: 60minsX 2 =120mins/week X 4 = 480 mins total dosage of intervention Participants also given a home exercise programme with a diary to record how long they practice for every day.
  Interventions: Other: Physiotherapy Core Stability Group Programme
- Clontarf Control Group 13-17 years (Active Comparator): Participants continue with usual care but do not include core stability or balance specific exercises in their physiotherapy programme for the duration of the control period. If they are receiving active physiotherapy treatment during this time, the duration, type and frequency of this intervention is recorded.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Physiotherapy Core Stability Group Programme — The aim of the intervention is to teach the participants active alignment and core stability, in order to influence their balance strategies. The exercises carried out will teach participants how and when to activate deep core stabilizing muscles. These exercises will be taught in a child-friendly way using imagery appropriate for the age of the participants. They will carry out activities like wall squats, 4-point kneeling, Transverses abdominis activation and gym ball sitting.
  Participants will also be supplied with a Home Exercise Programme (HEP) sheet with explanations for exercises that they will be asked to carry out on their 'off' days over the 4 week period. They will be asked to keep a record of their compliance with this.
  Arms: Clontarf Intervention Group 13-17 years; Intervention Group 7-12 years
Other: Control Group — The control group will partake in their usual physiotherapy care during the 4 week control period. They will not include core stability or balance specific exercises in their physiotherapy programme for the duration of the control period. If they are receiving active physiotherapy treatment during this time, the duration and frequency of this intervention is recorded
  Arms: Clontarf Control Group 13-17 years; Control Group 7-12 years

SUMMARY:
This study aims to determine if participation in a core stability physiotherapy group programme can improve the balance of children with cerebral palsy. It is hypothesised that teaching the children how and when to activate their deep core stabilising muscles may help improve their body awareness and their ability to control their alignment and therefore positively affect their balance. Children with cerebral palsy from the ages of 7 to 17, who can walk independently, will be randomly selected to join either the control group or intervention group, after completion of their baseline balance assessments. Each group will be re-assessed after completion of their 4 week intervention or control period.

DETAILED DESCRIPTION:
Introduction

The 'Core Muscles' are defined as '29 pairs of muscles that support the lumbo-pelvic hip complex in order to stabilize the spine, pelvis and kinetic chain during functional movement'.

Core stability refers to the control, co-ordination and synergism required by the core muscles for the maintenance of functional stability and balance. The role the core musculature plays in movement and postural control is long established. The understanding that our core muscles work in a feed-forward manner, laying the foundation of distal limb movement, formed the basis for studies into the use of core stability training programmes, such as pilates, core control training and spinal stability training, for improved postural control and balance.

Literature is replete with studies investigating the use of core stability programmes for varied populations from the adult population for chronic back pain to elite athletes for injury prevention and performance.

Studies investigating its use in adults with postural control impairment due to upper motor neuron lesions (UMN) from Multiple Sclerosis and Stroke showed positive effects on balance and mobility. The randomised controlled trial, by Chung et al, looked at the effects of a 4 week core stability exercise class on Dynamic Balance and Gait Function of 16 stroke patients. It showed a significant improvement of Timed-Up-And-Go (TUG) scores from 33.06 +-18.39sec to 27.64+- 13.73 sec (p=0.057) in the intervention group. Gait velocity (from 44.83+- 18.83 cm/s to 58.91 +- 18.21 ; p=0.024) and cadence ( from 74.55+- 13.85 steps/min to 84.07 +- 14.00 steps/min ; p=0.041) also showed significant improvement in the intervention group. To date there are no studies investigating the use or potential benefit of specific core stability intervention in the Cerebral Palsy (CP) population.

CP describes a group of permanent disorders of the development of movement and posture, causing activity limitation, that are attributed to non- progressive disturbances that occurred in the developing fetal or infant brain. It has been suggested that poor postural control may underlie delays and deviations in motor skill acquisition and development observed in children with CP. Therefore, it is important that treatment of children with CP tries to improve postural control and the evidence suggesting postural control mechanisms in school-age children with CP are modifiable signifies that this goal is achievable.

Young children with CP have been shown to use excessive, non-reciprocal trunk and hip muscle activation during walking. It has been hypothesized that one reason for this may be their need to compensate for poor control of their core deep stabilising muscles, thus limiting their ability to control changes in their body's centre of mass (COM) during dynamic movements. To understand this further we must look closer at the different functions of the core muscles.

The core muscles can be separated into large-lever, superficial global muscles, including the rectus abdominis and psoas major, that function as primary movers and smaller, deep, local muscles, including the Transverse Abdominis and Internal oblique, that function as primary stabilisers. It is postulated that if the deep stabilisers are not adequately functioning, then postural control is assisted by secondary compensatory activation of other muscles that typically function as primary movers like the hip flexors, knee flexors and spinal extensors. When a primary mover is being used to compensate for deep stabilisers, it becomes less efficient in its role in mobilizing and posturally adjusting.

An ineffective deep stabilizing system also limits the ability of the body to maintain the joints in a position where muscles are at a mechanical advantage. This can have an added 'weakening' effect on muscles that are essential for postural control, like the gluteus medius, as it reduces their force-generating capacity.

The objectives of the study are:

1. To measure changes in performance on a series of static, anticipatory and reactive balance tasks using three dimensional motion analysis in children who participate in core stability (intervention group) compared to children who continue their usual care (control group).
2. To compare changes in functional balance tests of the intervention group to the control group
3. To analyse qualitative data from a post intervention questionnaire to determine the broader effects of the 'Core stability' group intervention on the child's real life function, participation and quality of life.

Selection Criteria

The study aims to investigate the effects of a treatment intervention on children with Cerebral Palsy (CP). It is best research practice to choose a homogenous group of participants for meaningful results. It has been shown that in relation to balance of ambulatory children with spastic CP, a functional classification system (Gross motor Function Classification System-GMFCS level) can be used to group children more homogenously than traditional classification by diagnosis. On this basis, it was decided to include children with GMFCS levels I and II. Ambulatory children with a GMFCS classification level III were excluded as most studies showed a large gap in balance abilities between levels II to III. This would lead to a much greater variance in the participant sample.The Central Remedial Clinic (CRC) database of clients attending Clondalkin or Clontarf physiotherapy services will be used to generate a list of clients aged 7 to 17, with spastic CP diplegia or hemiplegia GMFCs level I or II for each centre.

The study inclusion/exclusion criteria will then be applied to this list. The clients not meeting the inclusion criteria or those meeting the exclusion criteria will be removed. The remaining clients will be invited to participate in the study and a list will be generated of participants who agree.

The resulting list will be split into 2 separate age groups (Age 7-12 years and Age 13-17 years) and unique identifying numbers will be assigned to each client on the day of their initial baseline assessment.

The clients will be assessed in groups of a minimum of 6 and maximum of 12 and will be randomised according to the procedure detailed below.

Sample Size

The sample size was calculated in Stata IC 13 (StataCorp, Texas, USA) using step length as the primary outcome measure. A previous study comparing gait in CP and typically developing children over level and uneven ground found a mean difference of 9cm (standard deviation 9cm) in step length between groups (Malone et al 2014, submitted for publication). With a power of 0.9 and significance level of 0.05, a sample size of 22 in each group was derived, giving a total of 44. To allow for a 10% drop out, it was decided to enroll 48 participants to the study.

Randomisation

A randomisation procedure will be carried out by an individual blinded to both the treatment and assessment procedure. The unique identifying number of the individual and their group will be in-putted into an electronic randomisation tool. Group assignment will be known to the treating therapists but not to the assessing therapist to ensure a single-blind design.

The participants will be allocated based on randomisation to either Intervention (I) or control (C).

Statistical analysis

The primary research question is whether core stability classes improve movement and function in the intervention group (I) compared to the control group (C). Data will be plotted graphically and described in the first instance using means, medians, standard deviations. Normality will be assessed using the Shapiro Wilk test. Groups will be inspected for baseline comparability. Quantitative parametric data from movement analysis assessment will be compared for (I) and (C) groups using analysis of co-variance including baseline levels of the outcome and adjusting for any baseline imbalances. Non-normally distributed data, e.g. Functional Walk Test, will be compared using Poisson regression.

Statistical analysis will be performed with Stata IC 13. Statistical assistance will be available from the Department of Epidemiology in RCSI.

Ethical Approval

Ethical approval has been obtained from the CRC Ethics committee

Informed Consent A written explanation of the study and core control group will be provided for the parent/guardian and participant. The information will be presented in a manner that is easy to understand and outline the risks and benefits of the study clearly. Each parent and participant will be given the opportunity to ask questions in writing or verbally and the parent/guardian will then sign a consent form. Refusal to participate in the study will not affect the client's general physiotherapy care from the CRC in any way.

Participants The control group will not work on focused balance specific core stability work in physiotherapy over the four-week control period. They will receive all other usual physiotherapy care during this period. Participants who are initially assigned to the control group will then be offered to participate in a Core Stability group after the control period assessments are completed. Therefore, all study participants (intervention and Control groups) will be given the opportunity to avail of the 'Core Stability' physiotherapy group programme. Each group will have to attend the same number of assessments (1 pre assessment and 1 post assessment)

Data Collection and Protection All data collected from the study will be restricted to the circumstances listed on the signed consent form. The procedures in place in relation to data storage and processing in the Gait Laboratory and the Physiotherapy Department in the CRC will be followed. Identifying information will only be stored in the CRC secure server.

Potential Risks During the Balance assessment in the gait laboratory, markers will be placed on the skin with adhesive tape. Taking these off may cause very slight discomfort. To alleviate this adhesive removal spray can be used.

The gait lab balance assessment is designed to be a measure of dynamic balance. Therefore, participants will be asked to do some tasks that may be challenging to them. They will be supervised at all times when carrying out the assessment by the independent assessor. Stand by assistance will be provided if required for safety.

The 'Core Stability' physiotherapy group intervention programme may be both mentally and physically challenging for the participants. It will involve concentration and repetition of activities. The group will be carried out under the supervision of two paediatric senior physiotherapists who work regularly with this CP population. These physiotherapists will have a strong knowledge base of this population's physical limitations. They are also experienced in how to encourage and motivate paediatric clients to carry out challenging activities.

ELIGIBILITY:
Inclusion Criteria:

* Children with spastic Cerebral Palsy (CP)
* Ages 7 - 17 (inclusive)
* GMFCS I-II (Gross Motor Function Classification System)
* Diplegia, Hemiplegia
* Balance problems identified (Determined by primary PT's treating problem list and/or score on balance assessments in use)
* Parental Informed Consent
* Can follow verbal instructions and willing to participate in a group intervention setting

Exclusion Criteria:

* Recent surgery to lower limbs (within past year)
* Botulinum Toxin (BTX-A) or serial casting to lower limbs within the last 3 months (or planned for during intervention or control period)
* Completed a core stability training group within the previous year
* Neurological or orthopaedic conditions unrelated to CP
* Behavioural difficulties limiting ability to participate in groups
* Intellectual difficulty that would make it difficult to comprehend and cooperate with treatment and/or testing

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-04 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Changes in performance of a static balance task ( single leg stand) using three dimensional motion analysis | Baseline and up to 3 weeks post intervention/control 4 week period
  o Relationship of Centre of Mass to Centre of Pressure
Changes in performance of an anticipatory balance task using three dimensional motion analysis | Baseline and up to 3 weeks post intervention/control 4 week period
  o Kinematic variables relating to trunk, pelvis, hip, knee and ankle movement at key points in the task of tandem walking.
Changes in stride length when balance is challenged during gait using three dimensional gait analysis | Baseline and up to 3 weeks post intervention/control 4 week period
  o Temporal-spatial parameters of stride length while walking over a 'wobbly road'. ( In gait lab setting this is achieved using bean bags placed under a mat.

SECONDARY OUTCOMES:
Changes in a series of functional Balance tests: Berg Balance Scale and Functional Walk Test | Baseline and up to 3 weeks post intervention/control 4 week period
Qualitative data from a post intervention questionnaire to determine the broader effects of the 'Core stability' group intervention on the child's real life function, participation and quality of life. | Up to 1 year Post intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Dara Dr Meldrum, BSc,MSc,PhD, Study Chair — Royal College of Surgeons, Ireland
Locations (1):
- Central Remedial Clinic, Dublin, Dublin, Ireland

REFERENCES:
- [Background] Anttila H, Autti-Ramo I, Suoranta J, Makela M, Malmivaara A. Effectiveness of physical therapy interventions for children with cerebral palsy: a systematic review. BMC Pediatr. 2008 Apr 24;8:14. doi: 10.1186/1471-2431-8-14. PMID 18435840
- [Background] Bar-Haim S, Al-Jarrah MD, Nammourah I, Harries N. Mechanical efficiency and balance in adolescents and young adults with cerebral palsy. Gait Posture. 2013 Sep;38(4):668-73. doi: 10.1016/j.gaitpost.2013.02.018. Epub 2013 Mar 21. PMID 23522668
- [Background] Chung EJ, Kim JH, Lee BH. The effects of core stabilization exercise on dynamic balance and gait function in stroke patients. J Phys Ther Sci. 2013 Jul;25(7):803-6. doi: 10.1589/jpts.25.803. Epub 2013 Aug 20. PMID 24259857
- [Background] Freeman JA, Gear M, Pauli A, Cowan P, Finnigan C, Hunter H, Mobberley C, Nock A, Sims R, Thain J. The effect of core stability training on balance and mobility in ambulant individuals with multiple sclerosis: a multi-centre series of single case studies. Mult Scler. 2010 Nov;16(11):1377-84. doi: 10.1177/1352458510378126. Epub 2010 Aug 10. PMID 20699285
- [Background] Gan SM, Tung LC, Tang YH, Wang CH. Psychometric properties of functional balance assessment in children with cerebral palsy. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):745-53. doi: 10.1177/1545968308316474. Epub 2008 Jul 21. PMID 18645187
- [Background] Hodges PW, Richardson CA. Feedforward contraction of transversus abdominis is not influenced by the direction of arm movement. Exp Brain Res. 1997 Apr;114(2):362-70. doi: 10.1007/pl00005644. PMID 9166925
- [Background] Hodges PW, Richardson CA. Transversus abdominis and the superficial abdominal muscles are controlled independently in a postural task. Neurosci Lett. 1999 Apr 16;265(2):91-4. doi: 10.1016/s0304-3940(99)00216-5. PMID 10327176
- [Background] Liao HF, Hwang AW. Relations of balance function and gross motor ability for children with cerebral palsy. Percept Mot Skills. 2003 Jun;96(3 Pt 2):1173-84. doi: 10.2466/pms.2003.96.3c.1173. PMID 12929770
- [Background] Liao HF, Mao PJ, Hwang AW. Test-retest reliability of balance tests in children with cerebral palsy. Dev Med Child Neurol. 2001 Mar;43(3):180-6. PMID 11263688
- [Background] Okada T, Huxel KC, Nesser TW. Relationship between core stability, functional movement, and performance. J Strength Cond Res. 2011 Jan;25(1):252-61. doi: 10.1519/JSC.0b013e3181b22b3e. PMID 20179652
- [Background] Prosser LA, Lee SC, VanSant AF, Barbe MF, Lauer RT. Trunk and hip muscle activation patterns are different during walking in young children with and without cerebral palsy. Phys Ther. 2010 Jul;90(7):986-97. doi: 10.2522/ptj.20090161. Epub 2010 Apr 29. PMID 20430948
- [Background] Quinn A, O'Regan M, Horgan F. Psychometric evaluation of the functional walking test for children with cerebral palsy. Disabil Rehabil. 2011;33(25-26):2397-403. doi: 10.3109/09638288.2011.573057. Epub 2011 Apr 20. PMID 21504407
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Shumway-Cook A, Hutchinson S, Kartin D, Price R, Woollacott M. Effect of balance training on recovery of stability in children with cerebral palsy. Dev Med Child Neurol. 2003 Sep;45(9):591-602. doi: 10.1017/s0012162203001099. PMID 12948326
- [Background] Woollacott M, Shumway-Cook A, Hutchinson S, Ciol M, Price R, Kartin D. Effect of balance training on muscle activity used in recovery of stability in children with cerebral palsy: a pilot study. Dev Med Child Neurol. 2005 Jul;47(7):455-61. doi: 10.1017/s0012162205000885. PMID 15991865
- [Background] Rydeard R, Leger A, Smith D. Pilates-based therapeutic exercise: effect on subjects with nonspecific chronic low back pain and functional disability: a randomized controlled trial. J Orthop Sports Phys Ther. 2006 Jul;36(7):472-84. doi: 10.2519/jospt.2006.2144. PMID 16881464
- [Background] Faries MD, Greenwood M. Core Training: Stabilizing the confusion. Strength and Conditioning Journal 29(2) :10-25, 2007
- [Background] Fredericson M, Moore T. Core Stabilization training for middle and long distance runners. New Stud. Athletics. 20:25-37, 2005.
- [Background] Hur JJ. Review of research on therapeutic interventions for children with cerebral palsy. Acta Neurol Scand. 1995 Jun;91(6):423-32. doi: 10.1111/j.1600-0404.1995.tb00441.x. PMID 7572035
- [Background] Malone A, Kiernan D, Saunders V, French H, O'Brien T. Do children with Cerebral Palsy change their gait over uneven ground? Proceedings of the Annual Meeting of the Clinical Movement Analysis Society UK and Ireland, 7-8 April 2014; Oswestry, Shropshire, UK.
- [Background] Kembhavi G, Darrah J, Magill-Evans J, Loomis J. Using the berg balance scale to distinguish balance abilities in children with cerebral palsy. Pediatr Phys Ther. 2002 Summer;14(2):92-9. doi: 10.1097/00001577-200214020-00005. PMID 17053689
- [Background] Williams EN, Carroll SG, Reddihough DS, Phillips BA, Galea MP. Investigation of the timed 'up & go' test in children. Dev Med Child Neurol. 2005 Aug;47(8):518-24. doi: 10.1017/s0012162205001027. PMID 16108451